CLINICAL TRIAL: NCT01364350
Title: TODAY2 Phase 1 Immediate Post-Intervention Observational Follow-up Study of the TODAY Clinical Trial Cohort
Brief Title: TODAY2 Phase 1 Immediate Post-Intervention Observational Follow-up Study
Acronym: T2P1
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kimberly, Principal Investigator of Coordinating Center, George Washington University
Other Study IDs: DK61230-T2P1
Record Dates: First submitted 2011-05-24; First posted 2011-06-02 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: type 2 diabetes mellitus; pediatrics; post-intervention study; metformin; complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine are collected on an annual basis and sent to the Central Biospecimen Laboratory for analysis and storage.
  Analyses performed on an annual basis are: HbA1c, insulin sensitivity and secreation (fasting glucose, insulin, C-peptide, and proinsulin), 2-hour OGTT, pancreatic autoimmunity, serum creatinine, liver function tests, lipids (LDL, triglycerides, free fatty acids, lipoprotein subclass levels, average LDL particle density, and total apoB levels), cardiovascular risk factors (fibrinogen, c-reactive protein, homocysteine vitamin B-12, plasminogran activator inhibitor-1, interleukin-6), microalbumin.
  HbA1c is also analyzed quarterly.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TODAY cohort: The cohort of participants diagnosed with type 2 diabetes ages 10 to <18 and obese at time of diagnosis who participated in the TODAY clinical trial are recruited, consented and followed.
  Interventions: Other: standard of care in general clinical practice

INTERVENTIONS:
Other: standard of care in general clinical practice — Participants consenting to receive study-provided care may be treated with metformin, insulin, statin, and ace-inhibitor, as needed for glycemic control and for comorbid conditions.

SUMMARY:
The purpose of this study is to continue to follow participants in the TODAY clinical trial as they transition to non-blinded, non-randomized standard diabetes care and management with monitoring and follow-up for up to 24 months (phase 1), during which time the TODAY data are analyzed and findings interpreted to develop a long-term observational protocol (phase 2). Data are collected during phase 1 for descriptive purposes; there is no primary hypothesis.

DETAILED DESCRIPTION:
TODAY (Treatment Options for type 2 Diabetes in Adolescents and Youth) was a multi-center study of the optimal approach to treatment of type 2 diabetes (T2D) in children and adolescents. The TODAY clinical trial of experimental interventions ended in February 2011. It is followed by TODAY2, a longitudinal study to continue the care and observation of the TODAY cohort beyond the end of the TODAY intervention trial. TODAY2 consists of two phases.

1. First is the immediate transition of TODAY participants to non-blinded, non-randomized standard diabetes care and management with monitoring and follow-up for up to 24 months. During this period, the findings of TODAY are analyzed and interpreted by the study group.
2. The second phase is a protocol for long-term longitudinal follow-up of the TODAY cohort, based on findings from TODAY.

The primary objective of the first phase of TODAY2 is to continue to follow the TODAY subjects for up to 24 months in order to begin to:

* understand the persistence of the effects of the different treatment regimens used in TODAY,
* describe the continued evolution of beta cell function, and
* describe the development of vascular complications and risk factors for complications.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the TODAY clinical trial.
* Provided informed consent to participate in T2P1.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: participants in the TODAY clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
effects of TODAY treatment assignment on long-term glycemic control | observed for 2 years in phase 1
  The primary objective of the first phase of TODAY2 is to begin to examine the persistence of effects of the TODAY treatment assignment on long-term glycemic control following discontinuation of randomized treatment. During this period, results of TODAY are produced and used to define additional outcomes for the second phase of TODAY2.

SECONDARY OUTCOMES:
glycemic control | observed for 2 years in phase 1
  HbA1c is the designated measure of glycemic control during T2P1. Mean HbA1c levels for participants from the three original TODAY treatment arms are compared as measures of the degree and durability of glycemic control after discontinuation of initial randomized therapy. The overall target is to maintain HbA1c levels as close to the normal range as possible in order to reduce long-term diabetes complications. TODAY2 continues to use HbA1c < 6% as the target.
safety | observed for 2 years in phase 1
  In TODAY2, subjects are treated with approved medications, i.e., metformin and/or insulin. No specific abnormalities are expected to develop in this cohort, given the well-documented safety record of these agents. However, abnormalities in laboratory tests (hemoglobin/hematocrit, liver function tests, calculated creatinine clearance), episodes of severe hypoglycemia, and incidence of side effects (e.g., gastrointestinal complaints) are tracked.
insulin sensitivity and secretion | observed for 2 years in phase 1
  An important component of TODAY2 is to continue to monitor insulin sensitivity and secretion in the TODAY cohort after discontinuation of randomized therapy to determine (1) the evolution of changes in insulin secretion and sensitivity as participants emerge from puberty and enter young adulthood and (2) the effect of each of the initial therapies on the progression of changes in insulin sensitivity and secretion.
  Insulin sensitivity and secretion are determined with fasting glucose, insulin, C-peptide, and proinsulin levels, OGTT-based indices, HOMA, and QUICKI measured annually.
cardiovascular risk factors | observed for 2 years in phase 1
  Both traditional and non-traditional CVD risk factors are measured in the first phase of TODAY2 and assessed overall as well as compared across initial treatment arms. Blood pressure is measured at every visit and specimens drawn annually for repeated measurements of lipids (free fatty acids, lipoprotein subclass levels, average LDL particle density, and total apoB level), fibrinogen, c-reactive protein, plasminogen activator inhibitor-1, homocysteine (vitamin B-12 to evaluate homocysteine levels), and interleukin-6.
microvascular complications | observed for 2 years in phase 1
  Quantitation of microalbuminuria is performed by obtaining spot urine measurements of microalbumin/creatinine ratio at annual visits. Abnormal values are confirmed with two additional samples within three months; diagnosis of microalbuminuria is made as a result of two out of three positive tests. Creatinine clearance (by calculation) is determined at annual visits.
  The presence of peripheral neuropathy is evaluated using the Michigan Neuropathy Screening Instrument (MNSI) performed annually.

CONTACTS AND LOCATIONS:
Overall Officials: Silva Arslanian, MD, Principal Investigator — University of Pittsburgh; Sonia Caprio, MD, Principal Investigator — Yale University; Leona Cuttler, MD, Principal Investigator — CWRU Rainbow Babies and Children's Hospital; Ken Copeland, MD, Principal Investigator — University of Oklahoma Health Science Center; Mitch Geffner, MD, Principal Investigator — Children's Hospital Los Angeles; Robin Goland, MD, Principal Investigator — Columbia University Naomi Berrie Diabetes Center; Lorraine Katz, MD, Principal Investigator — Children's Hospital of Philadelphia; Lori Laffel, MD, Principal Investigator — Joslin Diabetes Center; Barbara Linder, MD PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Jane Lynch, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Siripoom McKay, MD, Principal Investigator — Baylor College of Medicine; David Nathan, MD, Principal Investigator — Massachusetts General Hospital; Sherida Tollefsen, MD, Principal Investigator — Saint Louis University Health Sciences Center; Ruth Weinstock, MD PhD, Principal Investigator — State University of New York - Upstate Medical University; Neil White, MD, Principal Investigator — Washington University School of Medicine; Phil Zeitler, MD PhD, Study Chair — University of Colorado, Denver; Kathryn Hirst, PhD, Principal Investigator — George Washington University
Locations (16):
- United States (16):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Colorado Denver, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - George Washington University Biostatistics Center, Rockville, Maryland
  - Massachusetts General Hospital Diabetes Center, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Background] TODAY Study Group. Postintervention Effects of Varying Treatment Arms on Glycemic Failure and beta-Cell Function in the TODAY Trial. Diabetes Care. 2021 Jan;44(1):75-80. doi: 10.2337/dc20-0622. Epub 2020 Nov 10. PMID 33290248
- [Derived] TODAY Study Group; Shah RD, Braffett BH, Tryggestad JB, Hughan KS, Dhaliwal R, Nadeau KJ, Levitt Katz LE, Gidding SS. Cardiovascular risk factor progression in adolescents and young adults with youth-onset type 2 diabetes. J Diabetes Complications. 2022 Mar;36(3):108123. doi: 10.1016/j.jdiacomp.2021.108123. Epub 2022 Jan 3. PMID 35123868
- [Derived] Trief PM, Uschner D, Tung M, Marcus MD, Rayas M, MacLeish S, Farrell R, Keady J, Chao L, Weinstock RS. Diabetes Distress in Young Adults With Youth-Onset Type 2 Diabetes: TODAY2 Study Results. Diabetes Care. 2022 Mar 1;45(3):529-537. doi: 10.2337/dc21-1689. PMID 35015056
- [Derived] TODAY Study Group; Bjornstad P, Drews KL, Caprio S, Gubitosi-Klug R, Nathan DM, Tesfaldet B, Tryggestad J, White NH, Zeitler P. Long-Term Complications in Youth-Onset Type 2 Diabetes. N Engl J Med. 2021 Jul 29;385(5):416-426. doi: 10.1056/NEJMoa2100165. PMID 34320286